CLINICAL TRIAL: NCT06739161
Title: A Phase II Randomized Controlled Trial of Sintilimab in Combination with Chemotherapy ± Local Treatment for Oligometastatic Esophagogastric Junction/Gastric Adenocarcinoma
Brief Title: Sintilimab in Combination with Chemotherapy ± Local Treatment for Om-G/GEJ
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu Cancer Institute & Hospital (Other)
Responsible Party: Principal Investigator, Cheng Chen, Principal Investigator, Jiangsu Cancer Institute & Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCIR for G/GEJ
Record Dates: First submitted 2024-12-02; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Gastroesophageal Junction Adenocarcinoma
MeSH Terms: interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sintilimab combined with chemotherapy and local treatment (Experimental): ①Chemotherapy: Regimen follows guideline-recommended first-line therapy for advanced gastric cancer.
  ②Sintilimab (200 mg) is administered with chemotherapy every 21 days. Maintenance immunotherapy continues for up to 1 year after chemotherapy.
  ③Local Treatment : Performed during cycles 3-8 of immunochemotherapy. Radiotherapy is preferred, using a combination of high- and low-dose fractionation, tailored to tumor location, size, and proximity to critical organs.
  Interventions: Radiation: Sintilimab combined with chemotherapy and local treatment
- Sintilimab combined with chemotherapy (Active Comparator): ①Chemotherapy: Regimen follows guideline-recommended first-line therapy for advanced gastric cancer.
  ②Sintilimab (200 mg) is administered with chemotherapy every 21 days. Maintenance immunotherapy continues for up to 1 year after chemotherapy.
  Interventions: Combination Product: Sintilimab combined with chemotherapy only

INTERVENTIONS:
Radiation: Sintilimab combined with chemotherapy and local treatment — Treatment Regimens
  ①Chemotherapy: Regimen follows guideline-recommended first-line therapy for advanced gastric cancer.
  ②Sintilimab (200 mg) is administered with chemotherapy every 21 days. Maintenance immunotherapy continues for up to 1 year after chemotherapy.
  ③Local Treatment: Performed during cycles 3-8 of immunochemotherapy. Radiotherapy is preferred, using a combination of high- and low-dose fractionation, tailored to tumor location, size, and proximity to critical organs.
  Alternative local treatments, such as radiofrequency ablation or surgery, may be used if suitable.
  Arms: Sintilimab combined with chemotherapy and local treatment
Combination Product: Sintilimab combined with chemotherapy only — Treatment Regimens ①Chemotherapy: Regimen follows guideline-recommended first-line therapy for advanced gastric cancer.
  ②Sintilimab (200 mg) is administered with chemotherapy every 21 days. Maintenance immunotherapy continues for up to 1 year after chemotherapy.
  Arms: Sintilimab combined with chemotherapy

SUMMARY:
Gastric cancer is one of the most common and deadly cancers globally, with poor prognosis. About 70% of patients are diagnosed at an advanced stage, and the median overall survival (OS) is only 3-4 months. Current treatments, including immune checkpoint inhibitors combined with chemotherapy, have slightly improved survival, but most patients still experience disease progression during treatment, and those with PD-L1 CPS ≤5 do not benefit from immunotherapy.

Local radiotherapy, as a palliative treatment, can alleviate symptoms like bleeding, dysphagia, and pain, improving quality of life. Studies show that it significantly improves progression-free survival and may extend overall survival when added to chemotherapy. Therefore, combining local radiotherapy with immunochemotherapy may offer additional survival benefits for patients with advanced gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed esophagogastric junction (EGJ)/gastric adenocarcinoma.
2. Oligometastatic disease diagnosed via CT, MRI, or PET/CT:≤3 extracranial organs involved, ≤5 total metastatic lesions, each ≤5 cm in diameter,Regional lymph nodes count as one station; distant nodes counted per station.
3. No progression after two cycles of immunochemotherapy.
4. Primary and metastatic lesions at diagnosis eligible for local treatment.
5. All metastatic lesions measurable per RECIST 1.1.
6. Adequate hematological function: Neutrophil count ≥ 1.5 × 109/L, Platelets ≥ 100 × 109/L and Hemoglobin ≥90g/L.
7. Adequate liver function: Total bilirubin ≤ 1.5 × upper limit of normal (ULN); AST (SGOT) and ALT (SGPT) < 2.5 × ULN in the absence of liver metastases, or < 5 × ULN in case of liver metastases. ALP ≤ 2.5 × upper limit of normal (ULN); ALB ≥30g/L.
8. Adequate renal function: Serum creatinine ≤ 1.5 x ULN, and creatinine clearance ≥ 60 ml/min.
9. Adequate coagulation function: INR/PT≤ 1.5 x ULN, aPTT≤ 1.5 x ULN.
10. No serious concomitant disease that will threaten the survival of patients to less than 5 years.
11. Male or female. Age ≥ 18 years and ≤80 years.
12. Written (signed) informed consent.
13. Good compliance with the study procedures, including lab and auxiliary examination and treatment.
14. Female patients should not be pregnant or breast feeding.

Exclusion Criteria:

1. Non-adenocarcinoma histology of gastric/esophagogastric junction tumors, such as squamous cell carcinoma or neuroendocrine carcinoma.
2. Esophagogastric junction/gastric adenocarcinoma with positive Her-2 status requiring anti-Her-2 treatment.
3. Uncontrolled meningeal or peritoneal metastasis.
4. Peripheral neuropathy of grade ≥2.
5. Poor nutritional status, BMI <18.5 kg/m², or PG-SGA score ≥9.
6. Underwent major surgery or suffered a severe injury within 4 weeks prior to the first dose of the investigational drug.
7. Presence of uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage.
8. Received any investigational drug within 4 weeks prior to the first dose of the study drug.
9. Required systemic treatment with corticosteroids (daily >10 mg prednisone equivalent) or other immunosuppressive agents within 2 weeks prior to the first dose of the investigational drug.
10. Received an anti-tumor vaccine or live vaccine within 4 weeks before the first dose of the study drug.
11. Diagnosed with any active autoimmune disease or a history of autoimmune diseases.
12. History of immunodeficiency, including a positive HIV test, any acquired or congenital immunodeficiency diseases, or a history of organ transplantation or allogeneic bone marrow transplantation.
13. Any condition within 14 days prior to treatment requiring systemic corticosteroid therapy (dose>10mg/day of prednisone or equivalent) or other immunosuppressive treatments.
14. Presence of uncontrolled cardiac symptoms or conditions, such as:

    * NYHA Class II or higher heart failure
    * Unstable angina
    * Myocardial infarction within the past year
    * Clinically significant supraventricular or ventricular arrhythmias requiring clinical intervention.
15. Severe infection within 4 weeks prior to the first dose, including pneumonia requiring hospitalization, bacteremia, or infectious complications.
16. History of interstitial lung disease, non-infectious pneumonia, pulmonary fibrosis, or other uncontrolled acute pulmonary diseases.
17. Active pulmonary tuberculosis infection diagnosed by history or CT scan, or a history of active tuberculosis infection within the past year, or a history of untreated active tuberculosis infection more than one year ago.
18. Active hepatitis B or hepatitis C.
19. Laboratory abnormalities of sodium, potassium, or calcium greater than Grade 1 within 2 weeks before enrollment that cannot be corrected with treatment.
20. Known allergy to monoclonal antibodies, any PD-1 components, paclitaxel, capecitabine, or any components used in their formulations.
21. Pregnant or breastfeeding women, or women of childbearing potential who are unwilling or unable to use effective contraception.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-12-02 (Actual); Primary Completion 2027-12-02 (Estimated); Study Completion 2028-12-02 (Estimated)

PRIMARY OUTCOMES:
Progression free survival, defined as the time from randomization to disease progression or death, whichever occurs first. | From the date of randomization until tumor progression or death from any cause, whichever occurs first, assessed up to 24 months
  Progression will be assessed based on imaging studies and clinical evaluation, using RECIST v1.1 criteria. Data will be summarized using Kaplan-Meier estimates, and hazard ratios will be calculated.

SECONDARY OUTCOMES:
Overall Survival, defined as the time from randomization to death from any cause. | From the date of randomization until death from any cause, assessed up to 36 months
  Overall Survival will be assessed using Kaplan-Meier estimates and compared between groups using a log-rank test. Median survival and survival rates at specific time points will be reported.
Objective Response Rate, defined as the proportion of participants achieving a complete or partial response, as assessed by RECIST v1.1 criteria. | From the date of randomization until the date of first documented objective response, assessed up to 12 months
  Responses will be evaluated through imaging and clinical assessments, with data reported as a percentage along with corresponding 95% confidence intervals.
Time to Progression, defined as the time from randomization to the first documented disease progression, as assessed by RECIST v1.1 criteria. | From the date of randomization until the date of first documented progression, assessed up to 24 months
  Time to Progression will exclude cases of death that occur without documented disease progression. Kaplan-Meier estimates will be used for analysis.
Treatment Safety: Number of participants with treatment-related adverse events, as assessed by CTCAE v5.0. | From the date of randomization until the end of treatment, assessed up to 18 months
  Treatment-related adverse events will be categorized based on their severity and relationship to treatment, with descriptive statistics used to summarize their frequency and types.
Time to Symptom Deterioration, based on patient-reported outcomes using validated quality of life instruments (e.g., EORTC QLQ-C30). | From the date of randomization until the first documented symptom deterioration, assessed up to 12 months
  Time to Symptom Deterioration is defined as the time from randomization to the first clinically meaningful deterioration in symptom scores, determined by a predefined threshold. Kaplan-Meier methods will be used to analyze the data.

CONTACTS AND LOCATIONS:
Overall Officials: Cheng Chen, Principal Investigator — Jiangsu Cancer Institute & Hospital
Locations (1):
- ChengChen, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No